CLINICAL TRIAL: NCT02666391
Title: Safety and Exploratory Efficacy Study of UCMSCs in Patients With Ischemic Heart Disease (SEESUPIHD)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: South China Research Center for Stem Cell and Regenerative Medicine (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCMSC-2; NCT02568956 (obsolete NCT alias)
Record Dates: First submitted 2016-01-21; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Acute Myocardial Infarction; Myocardial Infarction; Ischemic Cardiomyopathy
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UCMSCs (Experimental): Intracoronary infusion of umbilical cord mesenchymal stem cells (UCMSCs)
  Interventions: Biological: umbilical cord mesenchymal stem cells
- controls (No Intervention): Standard medical treatment without umbilical cord mesenchymal stem cells (UCMSCs) infusion

INTERVENTIONS:
Biological: umbilical cord mesenchymal stem cells
  Arms: UCMSCs

SUMMARY:
The purpose of the present study is to evaluate the safety and exploratory efficacy of the umbilical cord mesenchymal stem cells for patients with ischemic heart diseases.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Ischemic cardiomyopathy caused by acute occlusion or severe stenosis of anterior descending artery;
* LVEF (left ventricular ejection fraction): 25-45%;
* Age between 18 and 70, borh gender;
* Women of childbearing age agreed to take contraceptive measures during the whole study period;
* No psychiatric illnesses and speaking dysfunction;
* Informed consent.

Exclusion Criteria:

* Structural heart disease, Valvular heart disease, Refractory hypertension(Unstable blood pressure control), LVEF<24%;
* Serious primary diseases of the liver, kidney and hematopoietic system, Abnormal liver function(glutamic-pyruvic transaminase(ALT), glutamic-oxaloacetic transaminase (AST) is 2 times higher than the normal value), creatinine(Cr) is higher than the upper limit of the normal value;
* Patients suffered from severe arrhythmia;
* Patients suffered from stent thrombosis;
* Patients receiving immunosuppressive therapy;
* Patients have tumor or other lethal diseases (expectation of life<6 months);
* Women who plan to be pregnant or are pregnant or nursing;
* Allergic constitution(Allergic to more than two kinds of drugs,food, or pollen);
* Other clinical trial participants within 3 months;
* Investigators judge other conditions not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in global left ventricular ejection fraction (LVEF)measured by echocardiography. | 1 week, 6 month, 12 month,18 month
Change in infarct size and myocardial viability within the infarcted region measured by emission computed tomography (ECT). | 1 week, 18 month

SECONDARY OUTCOMES:
Pump failure Killip classification | baseline, 1 week, 1 month, 6 month, 12 month,18 month
New York Heart Association(NYHA) classification | 1 week, 1 month, 6 month, 12 month,18 month
Occurrence of major adverse event | 3 day, 1 week, 1 month, 6 month, 12 month,18 month

REFERENCES:
- [Background] Gao LR, Pei XT, Ding QA, Chen Y, Zhang NK, Chen HY, Wang ZG, Wang YF, Zhu ZM, Li TC, Liu HL, Tong ZC, Yang Y, Nan X, Guo F, Shen JL, Shen YH, Zhang JJ, Fei YX, Xu HT, Wang LH, Tian HT, Liu DQ, Yang Y. A critical challenge: dosage-related efficacy and acute complication intracoronary injection of autologous bone marrow mesenchymal stem cells in acute myocardial infarction. Int J Cardiol. 2013 Oct 9;168(4):3191-9. doi: 10.1016/j.ijcard.2013.04.112. Epub 2013 May 4. PMID 23651816